CLINICAL TRIAL: NCT00493688
Title: A Study to Determine Whether Perioperative Energy Dynamics Correlates With Postoperative Outcomes
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0303; NCI-2024-06349 (Other: Clinicl Trials Reporting Program (CTRP))
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Cancer; Pelvic Cancer
Keywords: Abdominal Cancer; Pelvic Cancer; Perioperative Energy Dynamics; Cardiopulmonary Exercise Testing; CPET
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiopulmonary Exercise Testing (CPET)
  Interventions: Other: Cardiopulmonary Exercise Testing (CPET)

INTERVENTIONS:
Other: Cardiopulmonary Exercise Testing (CPET) — Pedaling on a Stationary Bicycle at 60 Revolutions Per Minute as the Resistance to Pedaling Gradually Increases.

SUMMARY:
To validate a new method for assessing perioperative risk in the cancer patient undergoing major cancer surgery.

In this proposed study researchers will:

1. Measure preoperative energy reserve capacity (fitness)
2. Determine if postoperative morbidity is a function of perioperative cardiopulmonary gas exchange metabolism

DETAILED DESCRIPTION:
Primary Objective:

• To characterize the effects of neoadjuvant therapy (chemotherapy, radiation therapy, and/or immunotherapy) on functional capacity in esophageal and lung cancer participants as measured by gas exchange parameters (%predicted AT, %predicted P-VO2, VO2 at AT & peak exercise, oxygen pulse, ΔVO2/ΔWR, ΔVE/ΔVCO2) obtained from CPET before and after neoadjuvant therapy.

Secondary Objectives:

• To characterize changes in CPET measures in participants treated with chemotherapy, radiation therapy, and/or immunotherapy followed by surgery and correlate these changes with postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age or older.
* Participants with newly diagnosed esophageal and lung cancer undergoing neoadjuvant chemotherapy, radiation therapy, and/or immunotherapy.
* Participants who have signed the consent form to participate in the study.
* Participants must have been evaluated in the Perioperative Evaluation and Management (POEM) Center or by a staff Anesthesiologist.
* All laboratory and diagnostic evaluations required or used to evaluate the patient must be completed. All participants must be approved to undergo anesthesia by the standards of the POEM Center.
* No samples belonging to vulnerable populations (children, pregnant women, cognitively impaired adults or prisoners) will be allowed from participation.

Exclusion Criteria:

* Participant is under age 18.
* Participant is unwilling to sign consent.
* Participant is unable to exercise (bedridden or wheel chair bound).
* Participant is enrolled in another study deemed by the investigator to affect oxygen metabolic efficiency and not presently the standard of care at MDACC.
* Participant's condition is deemed unsatisfactory for surgery after the preanesthetic evaluation.
* Participant has had a myocardial infarction within three months of the preanesthetic evaluation or presents with new or unstable angina.
* Participant has a history of a cerebrovascular accident or transit ischemic attacks within three months of the preanesthetic evaluation.
* Participant has a history of a pulmonary embolic event within three months of the preanesthetic evaluation.
* Participant is known to have acute or chronic deep vein thrombosis.
* Participant is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals scheduled for elective major intrabdominal surgery or pelvic surgeries surgeries (e.g. gastrectomy, esophagectomy, pancreatectomy, radical cystectomy, radical transabdominal debulking with or without intrabdominal hyperthermic perfusion, pelvic exenteration, retroperitoneal lymph node dissections, and low anterior resection).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-10-30 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Patient Perioperative Risk | Baseline + 30 days postoperatively monitoring for morbid events
  Measure preoperative energy reserve capacity (fitness) using perioperative energy dynamics where fitness is defined by gas exchange data during cardiopulmonary exercise testing as method of assessing perioperative risk

CONTACTS AND LOCATIONS:
Overall Officials: Anh Dang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org